CLINICAL TRIAL: NCT02849405
Title: Preliminary Evaluation of the Capacity of a Metabolic Hyperspectral Retinal Camera (MHRC) to Identify an Arteriosclerosis Spectral Signature in Retinal Arterioles
Brief Title: Evaluation of the Capacity of a Camera to Identify Signs of Arteriosclerosis in Retinal Arterioles
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jean-Claude Tardif (Other)
Collaborators: Montreal Heart Institute (Other); Polytechnique Montréal (Unknown)
Responsible Party: Sponsor-Investigator, Jean-Claude Tardif, Director, Research Center, Montreal Heart Institute
Organization: Montreal Heart Institute (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: ICM-ART-P
Record Dates: First submitted 2016-07-14; First posted 2016-07-29 (Estimated); Last update posted 2024-03-28 (Actual); Status verified 2024-03

CONDITIONS: Arteriosclerosis
MeSH Terms: conditions — Arteriosclerosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arteriosclerosis (Other): Hyperspectral camera for arteriosclerosis Diagnostic
  Interventions: Device: MHRC: Metabolic Hyperspectral Retinal Camera
- Healthy controls (Other): Hyperspectral camera for healthy control Diagnostic
  Interventions: Device: MHRC: Metabolic Hyperspectral Retinal Camera

INTERVENTIONS:
Device: MHRC: Metabolic Hyperspectral Retinal Camera — Comparison of hyperspectral signature of retinal arterioles between subjects suffering from arteriosclerosis and healthy control subjects.

SUMMARY:
Arteriosclerosis is a degenerative and dysmetabolic disease of the arterial walls. It is known to be the principal cause of coronary artery disease (CAD). Arteriosclerosis has an impact on the entire vascularization including the microvascularization. The retina is a nervous tissue that is supported by microvascularization. Therefore, systemic diseases that affect the nervous or the cardiovascular system are susceptible to have manifestations in the retina. Retinal signs associated to the risks to develop CAD (qualitative appreciation; diameter and appearance of arterioles) have been suggested. A quantitative approach would strengthen the interpretation of these evaluations.

The Metabolic Hyperspectral Retinal Camera (MHRC) - the experimental instrument - has the capacity to identify and quantify a variety of biomolecules specific to the retina and the optic nerve.

The purpose of this pilot study is to determine if the MHRC has the capacity to detect a specific hyperspectral signature in the retinal arterioles of subjects suffering from arteriosclerosis.

DETAILED DESCRIPTION:
In this pilot study, the main goal is to evaluate the capacity of the Metabolic Hyperspectral Retinal Camera (MHRC) - the experimental instrument - to identify the presence of a specific hyperspectral signature in the retinal arterioles of subjects suffering from arteriosclerosis while this signature should not be present in the retinal arterioles of control subjects considered healthy and without arteriosclerosis risk factors. The study is open, non-controlled and without randomization or placebo.

30 subjects of each group will be enrolled in the study for a total of 60 subjects. Recruitment will take place at the Montreal Heart Institute (Montreal, Quebec, Canada) and will be led by the research team of the Principal Investigator. Specific inclusion/exclusion criteria will differentiate subjects in each group. Once subjects fitting the inclusion/exclusion criteria will be identified, they will be enrolled and asked to sign the informed consent form approved by the Research Ethics and New Technology Development Committee (Montreal Heart Institute).

Following this step, an ophthalmic examination will be performed. During this examination, both eyes will be evaluated in order to detect the presence of eye pathologies (advanced cataracts, venous occlusion, age-related macular degeneration or glaucoma) that could interfere with the analysis of the MHRC optical imaging results. The ophthalmic examination consists first of a slit-lamp evaluation and secondly of an optic coherence tomography (OCT) plus a color image of the fundus (standard instruments commonly used in ophthalmology clinics) following the instillation of eye drops to dilate the pupils. The whole examination should last 45 minutes (it takes 15 to 20 minutes for the pupil to be sufficiently dilated to carry out the examinations). If the ophthalmic examination does not reveal any of the exclusion criteria, in the next minutes, the subject will be asked to undergo the baseline MHRC examination. This baseline imaging session will last a maximum of 15 minutes.

All data according to the light signal spectrum will be analyzed subsequently. Only depersonalized data, identified solely by the subject number, will be used by the investigators.

Risks associated to the subject's participation in this research project have been evaluated. Pupil dilation will be necessary to obtain quality images of the retina using conventional imaging techniques (OCT and fundus) and with the MHRC. The subject's pupils will remain dilated for 4 to 6 hours afterward, which may cause significant glare in areas where light is strong.. The MHRC is a research instrument which images the retina non-invasively and Health Canada authorization has been obtained for its use in the context of this study. The only foreseeable harm connected to its use is discomfort connected to the injection of light into the eye. The power of the monochromatic light source has been calculated to be well below the recommended exposure limits.. Very rigorous verifications were made according to the parameters fixed by the "American National Standard for safe use of laser" (ANSI 136.1) for laser radiation exposure.

Finally, all conflicts of interested are declared in the protocol and the informed consent form. Measures are in place to mitigate them in order to maintain research and data analysis integrity.

ELIGIBILITY:
Inclusion Criteria:

Subjects suffering from arteriosclerosis:

1. myocardial infarction
2. coronary angiography showing at least one coronary stenosis (more than 50%)
3. and/or coronary angioplasty
4. and/or coronary bypass.

Healthy control subjects:

1. absence of a medical history of cardiovascular disease
2. absence of medical history of cerebrovascular disease
3. absence of a medical history of peripheral arterial disease

Exclusion Criteria:

Healthy control subjects:

1. myocardial infarction or angina
2. known coronary stenosis
3. coronary angioplasty history or coronary bypass surgery
4. stroke or transient ischemic attack history
5. peripheral arterial disease history
6. active smoking or history smoking in the past 5 years
7. diabetes mellitus
8. familial hypercholesterolemia
9. poorly controlled hypertension (systolic blood pressure ≥150 mm Hg)

All subjects:

1. medium or high opacity of the lens (which interferes with the MHRC imaging)
2. bleeding in the vitreous (which interfere with MHRC imaging)
3. presence of venous occlusion, age-related macular degeneration or glaucoma
4. pupillary dilation inadequate or contra-indicated
5. deficient visual fixation
6. refractive error outside of the range -9 to +9
7. inability to obtain satisfactory images with the MHRC

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2016-12-21 (Actual); Primary Completion 2021-09-16 (Actual); Study Completion 2021-09-16 (Actual)

PRIMARY OUTCOMES:
Spectral intensity measures to visible and near infrared light around retinal arterioles in 30 patients with clearly defined atherosclerosis and 30 controls. | 1 Year
  Data will be aggregated for all arterioles identified in retinal image to produce a single outcome

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Claude Tardif, MD, Principal Investigator — Montreal Heart Insitute
Locations (1):
- Montreal Heart Institute, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Delori FC, Webb RH, Sliney DH; American National Standards Institute. Maximum permissible exposures for ocular safety (ANSI 2000), with emphasis on ophthalmic devices. J Opt Soc Am A Opt Image Sci Vis. 2007 May;24(5):1250-65. doi: 10.1364/josaa.24.001250. PMID 17429471
- [Background] Sliney D, Aron-Rosa D, DeLori F, Fankhauser F, Landry R, Mainster M, Marshall J, Rassow B, Stuck B, Trokel S, West TM, Wolffe M; International Commission on Non-Ionizing Radiation Protection. Adjustment of guidelines for exposure of the eye to optical radiation from ocular instruments: statement from a task group of the International Commission on Non-Ionizing Radiation Protection (ICNIRP). Appl Opt. 2005 Apr 10;44(11):2162-76. doi: 10.1364/ao.44.002162. PMID 15835362
- [Background] Hansson GK. Inflammation, atherosclerosis, and coronary artery disease. N Engl J Med. 2005 Apr 21;352(16):1685-95. doi: 10.1056/NEJMra043430. No abstract available. PMID 15843671
- [Background] Abramoff MD, Garvin MK, Sonka M. Retinal imaging and image analysis. IEEE Rev Biomed Eng. 2010;3:169-208. doi: 10.1109/RBME.2010.2084567. PMID 22275207
- [Background] Tabatabaee A, Asharin MR, Dehghan MH, Pourbehi MR, Nasiri-Ahmadabadi M, Assadi M. Retinal vessel abnormalities predict coronary artery diseases. Perfusion. 2013 May;28(3):232-7. doi: 10.1177/0267659112473173. Epub 2013 Jan 15. PMID 23322671
- [Background] Wong TY, Klein R, Sharrett AR, Duncan BB, Couper DJ, Tielsch JM, Klein BE, Hubbard LD. Retinal arteriolar narrowing and risk of coronary heart disease in men and women. The Atherosclerosis Risk in Communities Study. JAMA. 2002 Mar 6;287(9):1153-9. doi: 10.1001/jama.287.9.1153. PMID 11879113
- [Background] Patel SR, Flanagan JG, Shahidi AM, Sylvestre JP, Hudson C. A prototype hyperspectral system with a tunable laser source for retinal vessel imaging. Invest Ophthalmol Vis Sci. 2013 Aug 1;54(8):5163-8. doi: 10.1167/iovs.13-12124. PMID 23821191
- [Background] Shahidi AM, Patel SR, Flanagan JG, Hudson C. Regional variation in human retinal vessel oxygen saturation. Exp Eye Res. 2013 Aug;113:143-7. doi: 10.1016/j.exer.2013.06.001. Epub 2013 Jun 18. PMID 23791637
- [Background] Kang MH, Balaratnasingam C, Yu PK, Morgan WH, McAllister IL, Cringle SJ, Yu DY. Alterations to vascular endothelium in the optic nerve head in patients with vascular comorbidities. Exp Eye Res. 2013 Jun;111:50-60. doi: 10.1016/j.exer.2013.03.005. Epub 2013 Mar 19. PMID 23518407
- [Background] Koc S, Ozin B, Altin C, Altan Yaycioglu R, Aydinalp A, Muderrisoglu H. Evaluation of circulation disorder in coronary slow flow by fundus fluorescein angiography. Am J Cardiol. 2013 Jun 1;111(11):1552-6. doi: 10.1016/j.amjcard.2013.01.324. Epub 2013 Mar 25. PMID 23538021
- [Background] Sayin N, Kara N, Uzun F, Akturk IF. A quantitative evaluation of the posterior segment of the eye using spectral-domain optical coherence tomography in carotid artery stenosis: a pilot study. Ophthalmic Surg Lasers Imaging Retina. 2015 Feb;46(2):180-5. doi: 10.3928/23258160-20150213-20. PMID 25707042